CLINICAL TRIAL: NCT04278053
Title: Effects of Nitrosigine on Flow-Mediated Dilation Among Young Adults
Brief Title: Evaluation of Sports Supplements on Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Michelle Gray, Associate Professor - Exercise Science, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1812163576
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Determine the Effects of Nitrosigine and Citrulline-malate on Flow-mediated Dilation Among Young Adults
Keywords: flow-mediated dilation; vasodilation; Nitrosigine; Citrulline-Malate
MeSH Terms: conditions — Aneurysm | interventions — nitrosigine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, crossover design
Who Masked: Participant, Investigator
Masking Description: Both the participants and the researchers were blinded to the supplements until all data collection had been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitrosigine supplementation (Experimental): Ultrasound is a non-invasive way of determining the diameter of arteries. A total of 10 measurements will be taken of the brachial artery. After the initial 10 measurements (~3-5 minutes), flow-mediated dilation (FMD) was performed. Flow mediated dilation was performed with a Hokanson rapid cuff inflator. The cuff (blood pressure cuff) was position on the forearm (just above the wrist) and was inflated to 250-300mmHg for a period of 5 minutes to restrict blood flow. After the 5-minute inflation period, the cuff was deflated and vessel diameter was re-assessed (10 additional trails). Following the initial FMD assessment, Nitrosigine (1.5 g) was provided in an 8 ounce solution with a cherry flavoring to mask taste. After consumption, participants remained in ESRC for 60 minutes to allow for digestion of the substance. Following the 60-minute absorption period, FMD was re-assessed.
  Interventions: Dietary Supplement: inositol-stabilized arginine silicate
- Citrulline-Malate supplementation (Experimental): Ultrasound is a non-invasive way of determining the diameter of arteries. A total of 10 measurements will be taken of the brachial artery. After the initial 10 measurements (~3-5 minutes), flow-mediated dilation (FMD) was performed. Flow mediated dilation was performed with a Hokanson rapid cuff inflator. The cuff (blood pressure cuff) was position on the forearm (just above the wrist) and was inflated to 250-300mmHg for a period of 5 minutes to restrict blood flow. After the 5-minute inflation period, the cuff was deflated and vessel diameter was re-assessed (10 additional trails). Following the initial FMD assessment, Citrulline-Malate (8 g) was provided in an 8 ounce solution with a cherry flavoring to mask taste. After consumption, participants remained in ESRC for 60 minutes to allow for digestion of the substance. Following the 60-minute absorption period, FMD was re-assessed.
  Interventions: Dietary Supplement: inositol-stabilized arginine silicate
- Placebo (Placebo Comparator): Ultrasound is a non-invasive way of determining the diameter of arteries. A total of 10 measurements will be taken of the brachial artery. After the initial 10 measurements (~3-5 minutes), flow-mediated dilation (FMD) was performed. Flow mediated dilation was performed with a Hokanson rapid cuff inflator. The cuff (blood pressure cuff) was position on the forearm (just above the wrist) and was inflated to 250-300mmHg for a period of 5 minutes to restrict blood flow. After the 5-minute inflation period, the cuff was deflated and vessel diameter was re-assessed (10 additional trails). Following the initial FMD assessment, dextrose (8 g) was provided in an 8 ounce solution with a cherry flavoring to mask taste. After consumption, participants remained in ESRC for 60 minutes to allow for digestion of the substance. Following the 60-minute absorption period, FMD was re-assessed.
  Interventions: Dietary Supplement: inositol-stabilized arginine silicate

INTERVENTIONS:
Dietary Supplement: inositol-stabilized arginine silicate — Participants were asked to complete the experimental protocol in a 2-hour fasted state. Each participant's brachial artery FMD was assessed twice during each trial, once before supplement ingestion, and again 60 minutes post-ingestion. Male participants were required to wait for a minimum of seven days between trials as a supplement washout period. Female participants reported for supplement trials outside of their follicular phase of the menstrual cycle so that results were not confounded by changes in serum estradiol, which can significantly attenuate flow-mediated dilation. Sixty minutes after supplement consumption, each participant was asked which supplement they thought they had consumed. Participants were also asked whether they experienced any adverse side effects.

SUMMARY:
Many athletes seek to increase their plasma (blood) nitric oxide content prior to exercise in order to augment vasodilation. Increased vasodilation during exercise, especially high intensity resistance training, allows for more blood flow to muscle tissues, which may give the athlete benefits such as increased work capacity and acute muscle hyperemia, which is commonly referred to as muscle pump. Pre-workout supplements are typically taken 30 minutes to 1 hour prior to the onset of exercise, so the current investigation seeks to determine if citrulline malate or nitrosigine can effect vasodilation within 1 hour of supplementation, and if so, which supplement is more effective. Based on previous findings, we hypothesize that a certain exercise intensity needs to be present for citrulline malate and nitrosigine to have an effect, so a change may not be observable at rest.

DETAILED DESCRIPTION:
Data collection will be conducted by qualified research staff and students at the University of Arkansas Exercise Science Research Center (ESRC). Upon contact with the research team, a medical/health questionnaire will be sent via email to the subject. This will be the initial screening tool to determine if the subject qualifies for the project. The subjects must meet the inclusion and none of the exclusion criteria in order to qualify for the study. Participants will be instructed to do the following the day of data collection: 1. No caffeine, stimulants, or blood thinners (such as ibuprofen, advil, aspirin, warfarin, clopidogrel, etc.) 24 hours prior to testing. 2. Wear comfortable clothes (short sleeve top). 3. Take all medication as normal (aside from those mentioned in #1). Participant testing will be conducted as follows: participant arrives at ESRC; height, weight, blood pressure, and complete questionnaires (electronically): medical history, 24-hour dietary recall, International Physical Activity Questionnaire (IPAQ). IPAQ is a standardized questionnaire used to evaluate an individual's level of physical activity in their daily life. After completing all surveys, the subject will be asked to lie in a supine position for 15 minutes, then they will have the diameter of the brachial artery (medial side of upper arm) assessed with ultrasound (GE Logiq e). Ultrasound is a non-invasive way of determining the diameter of arteries. A total of 10 measurements will be taken of the brachial artery. After the initial 10 measurements (~3-5 minutes), flow-mediated dilation (FMD) will be performed. Flow mediated dilation will be performed with a Hokanson rapid cuff inflator. The cuff (blood pressure cuff) will be position on the forearm (just above the wrist) and will be inflated to 250-300mmHg for a period of 5 minutes to restrict blood flow. After the 5-minute inflation period, the cuff will deflate and vessel diameter will be re-assessed (10 additional trails). Following the initial FMD assessment, one of three supplements will be consumed: citrulline-malate (8 g), Nitrosigine (1.5 g), or placebo (8 g Dextrose). After consumption, participants will remain in ESRC for 60 minutes to allow for digestion of the substance. Following the 60-minute absorption period, FMD will be re-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, regularly exercising young adults

Exclusion Criteria:

* hypertension, metabolic disorders, previous consumption of pre-workout supplements 6 months prior to study, prescriptions medications known to effect the vasodilatory response.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Vasodilation | 60 minutes
  Amount of brachial vasodilation caused by supplementation as measured by flow-mediated dilation and ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gray, Ph.D, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No